CLINICAL TRIAL: NCT02691221
Title: ReliefLink: A Preventative Mobile Toolkit for Follow-Up Care of Psychiatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Nadine Kaslow, PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00083066
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Suicide, Suicidal Ideation
Keywords: Suicidal behavior, Mobile Application, Mobile Health Tool
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants with previous suicide attempt or ideation (Other): Participants will complete daily tasks assigned for completion through a downloaded application on their mobile device and completing six 2-hour long outcome assessment sessions including rater-lead scales over the course of six months.
  Interventions: Behavioral: Relief Link Application Daily Tasks

INTERVENTIONS:
Behavioral: Relief Link Application Daily Tasks — Participants will complete daily mood tracking and completion of a minimum of one stress management activity per day. Relaxation exercises to choose from on the current version of RL are audio files (i.e., no visuals), and consist of: Guided Meditation, Energizing Breath, Guided Visualization for Relaxation, Progressive Relaxation, Mindfulness Meditation Body Scan, and Mindfulness of Breathing.

SUMMARY:
The purpose of this study is to increase use and availability, as well as assess the feasibility of the ReliefLink (RL) application for use in conjunction with standard care to promote psychological health and prevent suicidal behavior.

DETAILED DESCRIPTION:
The aims of this study of ReliefLink application are to determine the utility of ReliefLink self-reports of suicidal ideation, negative emotions, loneliness, subjective well-being, flourishing, mental toughness, positive emotions, learned optimism, resilience, and post-traumatic growth. Additional aims are to evaluate the impact of ReliefLink on perceived access to/usage of care and resources and to explore participant acceptance of ReliefLink as a technological support for standard treatment through human systems engineering of treatment plan adherence and user interview.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as patients seeking behavioral health treatment through the Grady Health System
* Speak English
* Sought inpatient and/or outpatient treatment with Grady Health System following a suicide attempt or ideation.
* Has personal access to a functioning iPhone and service plan.

Exclusion Criteria:

* Has significant cognitive impairments.
* Is actively psychotic or has an imminently life-threatening medical/psychiatric condition per provider evaluation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in scores on 6 item Columbia Suicide Severity Rating Scale Screener (C-SSRS) | Baseline, 6 Months
  A comprehensive, semi-structured interview measure that uniquely measures the full spectrum of suicidality including passive and active suicidal ideation, suicidal intent as well as suicidal behaviors. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." A higher number of "yes" responses indicated an increased degree of suicidal ideation.
Change in scores on 20-item Positive-Negative Affect Scale (PANAS) | Baseline, 6 Months
  Consists of 10 positively and 10 negatively valanced word items. Items are rated by the participant for the extent they are feeling this "right now" on a scale of 1- slightly or not at all through 5- extremely. Total scores can range from 10-50, with higher scores representing higher levels of positive effect and lower scores having negative effect.
Change in scores on 20-item R-UCLA Loneliness Scale | Baseline, 6 Months
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from 1 (Never) to 4 (Often). A higher score indicates an increased degree of loneliness.
Change in scores on 14-item Mental Health Continuum Short Form (MHC-SF) | Baseline, 6 Months
  Consists of 14 items and measures the degree of emotional well-being as defined in terms of positive affect/satisfaction with life; social well-being, social acceptance, social actualization, social contribution, social coherence social integration, psychological well-being, personal growth, positive relations with others, purpose in life and self-acceptance. Choices for these items vary between 1 to 7. Individuals who exhibit low levels (i.e., 'never' or 'once or twice' during the past month) on at least one measure of hedonic well-being and low levels on at least six measures of positive functioning are diagnosed with languishing mental health.
Change in scores on 12-item Flourishing Scale (FS) | Baseline, 6 Months
  A measure of the participant's self-perceived success in relationships, self-esteem, purpose, and optimism. Items are rated on a seven point rating scale from 1 Strongly disagree to 7 Strongly agree. The scale provides a single psychological well-being score. A lower score indicates a decreased degree of well-being.
Change in scores on 8-item Grit-S scale | Baseline, 6 Months
  Measures the individual's tendency to sustain interest in and effort toward very long-term goals. Eight items are assessed using a Likert-like scale (1 = Not like me at all, 5 = Very much like me). There are two sub-scales: Perseverance of Effort and Consistency of Interests. A lower score indicates a decreased decreased levels of perseverance and passion for long-term goals.
Change in scores on 10-item Life Orientation Test - Revised | Baseline, 6 Months
  Measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 5-point scale (5 = I agree a lot, 1 = I DISagree a lot). A lower score indicates a decreased degree of life orientation.
Change in scores on 25-item Connor Davidson Resilience Inventory | Baseline, 6 Months
  Measures resilience. Range of scores (0-100). A score of 0 is suggestive of no resilience, a score of 100 is suggestive of high level of resilience.
Change in scores on 21-item Posttraumatic Growth Inventory | Baseline, 6 Months
  Self-reported measure of post-traumatic growth on a scale of 0 (Did not experience change as a result of their crisis) to 5 (experienced to a very great degree as a result of their crisis). A lower score indicates a decreased degree of posttraumatic growth.
11-item Effectiveness of Obtaining Resources scale (EOR) | 6 Months
  Calculates the mean of the effectiveness scores for obtaining resources from 11 different types of community resources including mental health treatment, church or clergy, health care, legal services, police, or social services.
Number of participants experiencing hospitalizations | 6 Months
  Number of hospitalizations self-reported by participants during semi-structured interview. No or infrequent hospitalizations would indicate successful support for the participant via the RL app.
Number of participants experiencing self-injury events | 6 Months
  Number of self-injury events reported during semi-structured interview. No or infrequent self-injury events would indicate successful support for the participant via the RL app.

SECONDARY OUTCOMES:
Number of participant reported barriers to care and resources | 16 Weeks
  The number of participant reported barriers to care and resources will be gathered through mobile phone internal usage data coded and a semi-structured interview. Acceptance of ReliefLink as a treatment resource would be suggested if there aren't significant reported barriers.
Participant adherence to assigned coping skills activities | 16 Weeks
  The frequency of Participant adherence to assigned coping skills activities will be gathered through mobile phone internal usage data coded and a semi-structured interview. Acceptance of ReliefLink as a treatment resource would be suggested if there was significant participant adherence.
Participant adherence to daily mood tracking | 16 Weeks
  The degree of Participant adherence to daily mood tracking will be gathered through mobile phone internal usage data coded and a semi-structured interview. Acceptance of ReliefLink as a treatment resource would be suggested if there is significant adherence to mood tracking.
Participant usage of resource location functions | 16 Weeks
  The frequency of Participant usage of resource location functions will be gathered through mobile phone internal usage data coded and a semi-structured interview. Acceptance of ReliefLink as a treatment resource would be suggested if is significant participant usage.
Participant positive feedback | 16 Weeks
  Participant positive feedback will be gathered through a semi-structured interview. Acceptance of ReliefLink as a treatment resource would be suggested if there is positive participant feedback received.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Kaslow, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No